CLINICAL TRIAL: NCT06711848
Title: A Comparative Analysis of the Effectiveness, Usability, Uptake, and Acceptability of an Educational Website and a Mobile Health Application Prototype in Improving Knowledge on Oral Cancer
Brief Title: Testing and Comparing the Impacts of Mhealth-Based and Web-Based Education on Oral Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rwanda (Other)
Collaborators: University of Peradeniya (Other); University of Ibadan (Other); Usmanu Danfodiyo University (Other); Saveetha University (Other)
Responsible Party: Principal Investigator, Kehinde Kazeem Kanmodi, Honorary Research Fellow, University of Rwanda
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: No 595/CMHS IRB/2024
Record Dates: First submitted 2024-11-18; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Oral Cancer; Health Education, Community; Digital Intervention; MHealth Application; MHealth Intervention
Keywords: mobile health; application; website; impact; knowledge; oral cancer; public health; intervention
MeSH Terms: conditions — Mouth Neoplasms; Health Education; Tooth, Impacted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (No Intervention): This is the control group (arm). No educational intervention on oral cancer will be administered to this group.
- Web-based Intervention Group (Experimental): A web-based educational intervention on oral cancer will be administered to this group.
  Interventions: Behavioral: A web-based educational intervention on oral cancer
- mHealth-based Intervention Group (Experimental): An app-based educational intervention on oral cancer will be administered to this group.
  Interventions: Behavioral: A mobile health app-based educational intervention on oral cancer

INTERVENTIONS:
Behavioral: A web-based educational intervention on oral cancer — This intervention will involve administering education, via a website, on the meaning, risks, clinical features, prevention, treatment, and supports on oral cancer.
  Arms: Web-based Intervention Group
Behavioral: A mobile health app-based educational intervention on oral cancer — This intervention will involve administering education, via a mhealth application prototype, on the meaning, risks, clinical features, prevention, treatment, and supports on oral cancer.
  Arms: mHealth-based Intervention Group

SUMMARY:
Introduction: Oral cancer is a malignant neoplastic disease affecting the lip, oral cavity (mouth) and/or the oropharynx. Despite the intense and diverse public health interventions on oral cancer prevention, the global prevalence rates of oral cancer and its major risk factors are still very high. Hence, oral cancer is an issue of serious global health importance.

Aim: To test and compare the effectiveness, usability, uptake, and acceptability of an educational website and a mobile health application prototype on oral cancer in improving oral cancer knowledge among university students.

Methods: This study will adopt a randomised control trial design, and it will be conducted among 75 first-year bachelor's degree students from five universities across two continents: University of Rwanda (Rwanda, Africa), Usmanu Danfodiyo University (Nigeria, Africa), University of Peradeniya (Sri Lanka, Asia), University of Ibadan (Nigeria), and Saveetha University (India, Aisa). The study participants will be in three groups (Group 1, Group 2, and Group 3). The participants in Group 1 will be the control group (n = 25 participants; 5 participants from each university); that is the group that will not receive an educational intervention. However, those in Group 2 (n = 25 participants; 5 participants from each university) will receive a web-based educational intervention on oral cancer while those in Group 3 (n = 25 participants; 5 participants from each university) will receive an app-based educational intervention on oral cancer. Pretest survey and posttest survey will be done for all participants. The data collected will be statistically analysed using the Statistical Package for Social Sciences (SPSS) version 28 software. Descriptive statistics will be done for all variables while inferential statistics (analysis of variance) will be done to test for associations between variables of interest.

Conclusion: The findings of this study will determine the effectiveness, usability, uptake, and acceptability of the tested digital intervention tools.

ELIGIBILITY:
Inclusion Criteria:

* being a first-year bachelor degree student of either University of Rwanda (Rwanda), University of Peradeniya (Sri Lanka), Usmanu Danfodiyo University (Nigeria), University of Ibadan (Nigeria), or Saveetha University (India)
* being within the age range of 18 to 39 years
* having a personal smartphone
* willingness to participate in the study

Exclusion Criteria:

* being a member of staff or a visitor or a non-first year bachelor degree student of University of Rwanda (Rwanda), University of Peradeniya (Sri Lanka), Usmanu Danfodiyo University (Nigeria), University of Ibadan (Nigeria), or Saveetha University (India)
* being a student of a tertiary institution not selected for the study
* being below the age of 18 years or above the age of 39 years.
* not having a personal smartphone
* not willing to participate in the study

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-01-05 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Measurement of change in baseline knowledge on oral cancer four weeks post-intervention using a questionnaire | From enrollment to the end of educational intervention at 4 weeks
  This primary outcome measure will be a change in knowledge on oral cancer at four weeks after the delivery of the intervention, and this will be done using a questionnaire. All participants in both the control and intervention groups will be evaluated at baseline and at endline.
  This outcome will be measured using a questionnaire. This questionnaire was developed by the investigators. The questionnaire will obtain assess the participants' knowledge of oral cancer through the use of 10 multiple choice questions

SECONDARY OUTCOMES:
Measurement of the usability of the intervention tools using an adapted version of the user Mobile Application Rating Scale | At the end of educational intervention at 4 weeks
  This secondary outcome measure will be on the usability of the intervention tools, and this will be done using a questionnaire. Only those participants in the intervention groups will be evaluated on this outcome, and this will be done at post-intervention survey stage.
  This outcome will be measured using a questionnaire. This questionnaire was adapted from a standardised instrument called the "user Mobile Application Rating Scale". This instrument uses diverse Likert scales with a Likert score of 1 representing the extreme negative outcome (lowest rating on the tool's usability) while a score of 5 representing the extreme positive outcome (highest rating on the tool's usability).
Measurement of the uptake of the intervention tools using an adapted version of the user Mobile Application Rating Scale | At the end of educational intervention at 4 weeks
  This secondary outcome measure will be on the uptake of the intervention tools, and this will be done using a questionnaire. Only those participants in the intervention groups will be evaluated on this outcome, and this will be done at post-intervention survey stage.
  This outcome will be measured using a questionnaire. This questionnaire was adapted from a standardised instrument called the "user Mobile Application Rating Scale". This instrument uses diverse Likert scales with a Likert score of 1 representing the extreme negative outcome (lowest rating on the tool's uptake) while a score of 5 representing the extreme positive outcome (highest rating on the tool's uptake)
Measurement of the acceptability of the intervention tools using an adapted version of the user Mobile Application Rating Scale | At the end of educational intervention at 4 weeks
  This secondary outcome measure will be on the acceptability of the intervention tools, and this will be done using a questionnaire. Only those participants in the intervention groups will be evaluated on this outcome, and this will be done at post-intervention survey stage.
  This outcome will be measured using a questionnaire. This questionnaire was adapted from a standardised instrument called the "user Mobile Application Rating Scale". This instrument uses diverse Likert scales with a Likert score of 1 representing the extreme negative outcome (lowest rating on the tool's acceptability) while a score of 5 representing the extreme positive outcome (highest rating on the tool's acceptability).

CONTACTS AND LOCATIONS:
Overall Officials: Kehinde Kanmodi, BDS, MPH, Principal Investigator — University of Rwanda; Peace Uwambaye, BSC, MPH, PhD, Study Director — University of Rwanda; Afeez Salami, BDS, Study Director — University of Ibadan; Bello Almu, BSC, MSc, MPP, Study Director — Usmanu Danfodiyo University; Karthikeyan Ramalingam, BDS, MDS, Study Director — Saveetha University; Yovanthi Jayasinghe, BSc, PGD, Study Director — University of Peradeniya; Timothy Aladelusi, BDS, MSc, Study Director — University of Ibadan; Akinyele Adisa, BDS, Study Director — University of Ibadan; Jimoh Amzat, BSC, MA, MSc, PhD, Study Director — Usmanu Danfodiyo University; Ruwan Jayasinghe, BDS, MSc, Principal Investigator — University of Peradeniya
Locations (5):
- Saveetha University, Tamil Nadu, India
- Nigeria (2):
  - University of Ibadan, Ibadan, Oyo State
  - Usmanu Danfodiyo University, Sokoto, Sokoto State
- University of Rwanda, Kigali, Kigali, Rwanda
- University of Peradeniya, Peradeniya, Sri Lanka

IPD SHARING:
Plan to Share IPD: Yes
The names, and any other personal information that could potentially identify the participants will not appear in any reports or publications. The participants will be assigned a unique study identifying number (or pseudonym) which will be recorded only on a link document. This link document will be stored separately on the U-drive from both the person identifiable consent forms and the pseudo-anonymised data. Any participant that wishes to withdraw would email the researcher without giving a reason. As soon as the last date allowed for withdrawal has passed the coding (link) document will be securely destroyed and the data rendered non-person identifiable. Withdrawal is not possible after this point.
  The consent form will be stored for up to 10 years on the U-drive of the principal investigators, separate to other study data, as it is an important document. This is in case other scientists wish to raise questions about the results that need checking again.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Start date: 05 June 2025 End date: 05 May 2035
Access Criteria: Only the anonymised IPD documents will be shared and such can be shared upon reasonable request.